CLINICAL TRIAL: NCT00389116
Title: Value of CT-Scan and Oral Gastrografin in the Management of Post Operative Small Bowel Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Scotté, Pr, CHU Rouen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2005/069/HP
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Small Bowel Obstruction
MeSH Terms: interventions — Diatrizoate Meglumine; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: gastrograffin
- 2 (Placebo Comparator)
  Interventions: Drug: water

INTERVENTIONS:
Drug: gastrograffin — ingestion
  Arms: 1
Drug: water — oral water ingestion
  Arms: 2

SUMMARY:
Small bowel obstructions are responsible for 2 to 5% of emergency hospital admissions and 20% of all emergency surgical procedures. In 60 to 80% of cases, acute small bowel obstructions are the consequence of intraperitoneal postoperative adhesions. They constitute an extremely frequent pathology, leading to a high rate of hospital admissions and money expense.

Management of small bowel obstruction is based on 2 options: either a surgical approach where all patients are operating on, or a conservative treatment in which surgery is proposed in case of failure of medical treatment. The surgical approach leads to operate on an excessive rate of patients while the medical approach increases the risk of increased small bowel resection, morbidity rate or hospitalization duration.

In order to improve the management of small bowel obstruction, it seems necessary to better distinguish patients that need an emergency surgical procedure from patients in which medical treatment will be useful. Many studies have been performed to investigate the value of imaging in the management of small bowel obstruction, using abdominal X-ray, oral gastrografin administration or CT-Scan.

The aim of this study is to analyse the effect of a systematic performance of imaging investigation on the management of patients presenting with a postoperative small bowel obstruction.

All patients suffering from a postoperative small bowel obstruction will be included in this study. They will be randomised in 2 groups. In group S, patients will have CT-Scan and oral water administration while in group SG, Patients will have CT-Scan and oral gastrografin administration The major end point of this study is to analyse whether imaging examination can reduce the need for a surgical approach or the rate of small bowel resection and to determine its influence on fasting time or hospitalization duration

ELIGIBILITY:
Inclusion Criteria:

* Small bowel obstruction in patients with previous abdominal surgery

Exclusion Criteria:

* Age less than 18 years
* Early small bowel obstruction (less than 4 weeks following abdominal surgery)
* Small bowel obstruction in the course of digestive cancer.
* Hyperthermic small bowel obstruction
* Small bowel ischemia (fever, peritoneal signs, increased leucocytosis)
* Pregnancy ( Elevated béta HCG levels)
* Inflammatory bowel disease
* Previous abdominal radiotherapy
* Pneumoperitoneum
* Colorectal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Need for surgical management | 2 months

SECONDARY OUTCOMES:
Sensibility and specificity of gastrografin oral administration | 2 months
Sensibility and specificity of CT-Scan. | 2 months
Sensibility and specificity of abdominal X-ray. | 2 months
Fasting time | 2 months
Hospitalization time | 2 months
Number of small bowel resection | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: michel scotté, MD,PhD, Principal Investigator — CHU Rouen; francois mauvais, MD, Study Director — chg Beauvais; jean-marc regimbeau, MD, PhD, Study Director — CHU amiens
Locations (1):
- CHU, Rouen, France

REFERENCES:
- [Derived] Cosse C, Regimbeau JM, Fuks D, Mauvais F, Scotte M. Serum procalcitonin for predicting the failure of conservative management and the need for bowel resection in patients with small bowel obstruction. J Am Coll Surg. 2013 May;216(5):997-1004. doi: 10.1016/j.jamcollsurg.2012.12.051. Epub 2013 Mar 19. PMID 23522439